CLINICAL TRIAL: NCT05506722
Title: The Using of the Testes' Shocker in Improving the Sperms' Activity and the Spermatogenesis Process Among Infertile Men
Brief Title: Using of Testes Shocker in Improving the Spermatogenesis and Sperms Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Doctor (MBChB), University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS2
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Infertility, Male; Infertility Unexplained; Infertility Due to Complete Spermatogenic Arrest; Oligospermia; Asthenozoospermia; Necrospermia
Keywords: Infertility; Testes shocker; Electric shocks
MeSH Terms: conditions — Infertility, Male; Oligospermia; Asthenozoospermia; Infertility

STUDY DESIGN:
Intervention Model Description: Double blinded two groups, one is the treated group and the other is the placebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: By mixing the devices together and giving them to the participants blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testes shocker (Active Comparator): This device is working and giving the electrical shocks regularly.
  Interventions: Device: Testes shocker
- Fake Testes shocker (Placebo Comparator): This device is not giving electricity but it is working with a red light, so the participants cannot suspect it.
  Interventions: Device: Testes shocker

INTERVENTIONS:
Device: Testes shocker — It is a device that give electric shocks (up to 5 milli Amperes) and it is designed to contain both the testes within it.

SUMMARY:
Infertility was reported in approximately 15% of all heterozygous couples, with male factor accounting for nearly half the cases. This typically occurs due to low sperm production, sperm dysfunction, and sperm delivery obstruction. Etiology of male infertility can be attributed to many factors including acute or chronic illness, accidents, and lifestyle choices.

DETAILED DESCRIPTION:
This study demonstrated that using a painless, convenient at-home device could significantly improve sperm motility and count. This device can be utilized to tackle (for unexplained infertility) the significant issue of infertility in a cost-effective, safe and efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Infertile male with oligosperma, necrospermia, asthenozoospermia or hypospermia. Must not taking any drugs or medications for infertility and has nit any congenital diseases in the genital tracts or chronic diseases.

Exclusion Criteria:

* Have congenial genital tract disease, has a chrome disease, has other than the above mentioned causes for infertility or taking medications that can affect the fertility.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only those who consider themselves as males and have males genital organs of penis and testes were included.
Enrollment: 250 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Semen analysis | 4 months
  By taking the semen from the participants at baseline and then after each month and analyse it.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Talib T Hashim, MBChB, Principal Investigator — University of Baghdad, College of Medicine
Locations (1):
- Al-Dar medical Center, Nasiriyah, Thi Qar, Iraq

IPD SHARING:
Plan to Share IPD: No